CLINICAL TRIAL: NCT04984954
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Shexiang Baoxin Pill on Coronary Microvascular Dysfunction
Brief Title: Evaluate the Efficacy and Safety of MUSK Pill on Coronary Microvascular Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMPE202001
Record Dates: First submitted 2021-07-04; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Angina Pectoris; Coronary Heart Disease; X Syndrome, Angina; Non Obstructive Coronary Artery Disease
Keywords: Shexiang Baoxin Pill; Musk pill; Patients with coronary microvascular dysfunction
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Microvascular Angina | interventions — musk

STUDY DESIGN:
Intervention Model Description: 1:1 stratified block random grouping according to the center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This is a multicenter, randomized, double-blind, placebo-controlled clinical trial. Patients were treated with the trial drug or placebo in a 1:1 ratio. The experimental group was treated with MUSK pill (4 pills / day, 3 times / day) on the basis of conventional treatment until the end of follow-up
  Interventions: Drug: MUSK pill
- Placebo group (Placebo Comparator): The control group was given placebo 4 capsules / day, 3 times / day, until the end of follow-up.
  Interventions: Drug: MUSK pill

INTERVENTIONS:
Drug: MUSK pill — This is a multicenter, randomized, double-blind, placebo-controlled clinical trial. Patients were treated with the trial drug or placebo in a 1:1 ratio. The experimental group was treated with MUSK pill (4 pills / day, 3 times / day) on the basis of conventional treatment until the end of follow-up
  Other Names: Placebo

SUMMARY:
Objective to evaluate the effect of Shexiang Baoxin Pill on myocardial ischemia in patients with coronary microvascular dysfunction (non obstructive coronary heart disease) through a randomized, double-blind, placebo-controlled clinical multicenter study.At the same time, the effects of exercise tolerance and quality of life were also observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80, male or female;
2. Selective coronary angiography or coronary CTA showed that the diameter of coronary artery ≥ 2.5mm, the degree of stenosis < 50%, without myocardial bridge;
3. They were able to perform treadmill exercise, and the treadmill test (EET) was positive;
4. Angina pectoris was found;
5. Patients are willing to follow up and sign informed consent; All the above criteria should be met.

Exclusion Criteria:

1. Coronary heart disease complicated with hypertrophic cardiomyopathy;
2. There was a history of AMI, PCI and CABG, and myocardial bridge was found by angiography or CTA;
3. Patients with severe medical diseases (liver, kidney, hematopoietic system and other serious primary diseases, etc.);
4. Mental disorders and mental diseases;
5. Patients with pulmonary failure and NYHA heart function grade III-IV, unable to carry out exercise test;
6. Contraindications of Shexiang Baoxin Pill: forbidden for pregnant women;
7. Those who have known history of allergy to Shexiang Baoxin Pills;
8. Recently, the patient has taken Shexiang Baoxin Pill and other anti ischemic traditional Chinese medicine regularly, or it contains borneol, toad venom and other ingredients in Shexiang Baoxin Pill;
9. Combined with frequent ventricular premature beats, ventricular tachycardia, atrial fibrillation, sinoatrial block, atrioventricular pathway block, left bundle branch block and right bundle branch block, which may affect the judgment of exercise ECG results;
10. Researchers think that there are other factors that are not suitable to participate in the trial; If one of the exclusion criteria is met, it can be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the difference of HRR between the experimental group and the placebo group was significant | At the end of treatment (8 weeks (± 1 week))
  Definition of abnormal heart rate recovery: peak HR during exercise - HR one minute into recovery at the end of exercise is defined as abnormal heart rate recovery when HR one minute into recovery is less than 12 beats / min.

CONTACTS AND LOCATIONS:
Overall Officials: HaiMing Shi, doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China